CLINICAL TRIAL: NCT01383811
Title: Clinical and Neuroendocrine/Metabolic Benefits of Exercise in Treatment Resistant Depression (TRD): A Feasibility Study
Brief Title: Exercise in Treatment Resistant Depression (TRD): A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Ravi Singareddy, Associate Proffesor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34749EP
Record Dates: First submitted 2011-06-23; First posted 2011-06-28 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Treatment Resistant Depression
Keywords: Treatment Resistant Depression; Exercise
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Motor Activity | interventions — Exercise; Waiting Lists; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate Intensity Aerobic Exercise (Active Comparator)
  Interventions: Other: Moderate Intensity Aerobic Exercise; Other: Wait-list
- Wait List/Usual Care (Other): The subjects in this group will continue to receive the usual treatment that they were on at the time of enrollment through the wait list period of 12 weeks. Subsequently they will receive the 12 weeks of aerobic exercise program intervention
  Interventions: Other: Wait-list

INTERVENTIONS:
Other: Moderate Intensity Aerobic Exercise — Individuals in this group will receive moderate intensity exercise in addition to their usual care (Medications+/-Psychotherapy). The moderate intensity exercise program will involve gradual progression in exercise intensity and duration. During the first 4 weeks, participants will attend 3 supervised sessions/week and will be asked to complete at least 2 unsupervised aerobic exercise sessions/week. From weeks 5-8 the number of supervised sessions will be 2/week with at least 3 unsupervised aerobic exercise sessions/week. From weeks 9-12, the participants will have only 1 supervised session/week and will be asked to complete at least 4 unsupervised aerobic exercise sessions/week. In total, the participants will be required to complete 150 minutes of moderate physical activity/week.
  Other Names: Exercise; Aerobic Exercise
  Arms: Moderate Intensity Aerobic Exercise
Other: Wait-list — The wait list/usual care group will continue with their usual standard treatment (Medications +/- Psychotherapy) as before.
  Other Names: Usual care; Care as usual; Standard Care

SUMMARY:
The objective of this study is to determine the effects of adjunct exercise in treatment resistant depression. The central hypothesis for the research is that adjunct exercise with usual care in Treatment Resistant Depression (TRD) will have significant effects in improving the psychiatric symptoms in comparison to usual care alone.

DETAILED DESCRIPTION:
Participants with treatment resistant depression will be recruited to participate in a 12-week clinical trial on the effects of adjunct moderate-intensity exercise versus usual care. Primary outcome measure will be reduction in baseline scores on Hamilton Depression Rating Scale (17 item). Secondary outcome measure will include reduction in baseline scores of clinical global impression severity, pittsburgh sleep quality index global score, scores on beck depression inventory, and improvement in actigraphic sleep.

ELIGIBILITY:
Inclusion Criteria:

* Being sedentary (exercising less than 3 times/week for > 20 minutes at moderate/vigorous intensity for each bout)
* Ability to come for supervised exercises up to 5 days/week.
* On stable doses of medication or psychotherapy (within last 1 month) for underlying depression and willingness to continue on stable dose or therapy schedule during active phase of study participation, with the exception of during acute exacerbation of symptoms of psychiatric illness.
* Being able to read, understand, and provide written informed consent.

Exclusion Criteria:

* DSM-IV TR Axis I diagnosis of bipolar disorder, schizophrenia or schizophrenia spectrum disorder, or substance or alcohol abuse/dependence disorder (except nicotine dependence) in the past 12 months. Patients with current primary anxiety disorder will also be excluded.
* Behavioral or personality disturbances, which may significantly interfere with study participation.
* Evidence of acute suicidal risk.
* Medical contraindication for physical exercise (significant orthopedic or cardiopulmonary disorder) that would prevent regular aerobic exercise. The American College of Sports Medicine criteria for risk stratification will be used and where indicated medical clearance for exercise will be obtained through the subject's primary care physician.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline on Hamilton Rating Scale for Depression-17 item (HRSD17)score | Baseline, 6 weeks, and 12 weeks
  Hamilton Rating Scale for Depression-17 item (HRSD17, a well standardized measure of depression will be the primary measures of efficacy.

SECONDARY OUTCOMES:
Reduction in baseline scores of clinical global impression severity | Baseline, 6 weeks, and 12 weeks
Change from baseline on Beck Depression Inventory-II score | Baseline, 6 weeks, 12 weeks
  This is a widely used reliable and standardized measure of depression.
Change from baseline on Pittsburgh Sleep Quality Index (PSQI) global sleep quality score | baseline, 6 weeks, 12 weeks.
  PSQI is a widely used, reliable and standardized measure of subjecitve sleep

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Singareddy, MD, Principal Investigator — Penn State Univ. College of Medicine
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States